CLINICAL TRIAL: NCT02760706
Title: Preliminary Assessment of the Added Diagnostic Value of Dual Energy Computed Tomography (DECT) Images Using Data Acquired on a Spectral Detector Computed Tomography (SDCT)
Brief Title: Preliminary Assessment of Added Diagnostic Value of Dual Energy CT Images Using Data Acquired on a Spectral Detector CT
Status: Completed | Type: Observational
Sponsor: Philips Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: SDCTUH08-13-12
Record Dates: First submitted 2013-11-24; First posted 2016-05-04 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Compare Image Quality Between SDCT and Conventional CT Images of Any Tissue Lesion, Determine Optimal Monochromatic Energy Level for a Coronary Artery Image
MeSH Terms: interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Computed Tomography scan

SUMMARY:
Study hypothesis: Post-processed SDCT images provide additional diagnostic value over conventional CT datasets.

The CT examination would be a clinically-necessary, standard-of-care CT performed as per the clinical indication. The protocol and scan parameters for the CT exam will be similar to that of an equivalent scan performed with any other CT scanner. There would be no additional scanner of injection of any drug specifically for the study. The conventional CT images generated by the scanner will be used for clinical purposes as routinely practiced.

ELIGIBILITY:
Inclusion Criteria:

* a patient scheduled for a clinically indicated CT scan for one or more of the following body regions/organ systems:
* head and neck
* body (chest and abdomen/pelvis)
* cardiovascular structures.
* these scans may be without contrast, with contrast enhancement, or CT angiograms.

Exclusion Criteria:

* under the age of 18 years old
* standard exclusion criteria for CT scans

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring a clinically-necessary CT scan
Sampling Method: Non-Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2013-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Determine if Post-processed SDCT images provide additional diagnostic value over conventional CT datasets. | 6 months
  Data will be recorded as mean +/- standard deviation for each parameter. Student's t test and Wilcoxon's test will be performed to compare objective and subjective data respectively. In addition, differences on lesion detection and characterization, sensitivity, specificity and accuracy of conventional CT and SDCT images will be compared using a receiver operating curve (ROC) analysis. Additionally, agreement between both readers will be evaluated using Cohen´s kappa test (poor agreement for κ ≤ 0.19; fair agreement for κ = 0.2-0.39; moderate agreement for κ = 0.4-0.59, substantial agreement for κ = 0.6-0.79 and very good agreement for κ = 0.8-1.00; 19). A P value of <0.05 will be required for statistical significant difference.

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Gilkeson,, M.D., Principal Investigator — University Hospitals Cleveland Medical Center; Prabhakar Rajiah,, M.D., Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States